CLINICAL TRIAL: NCT02311569
Title: Effects of Sympathicomimetic Agonists on the Disease Course and Mutant Allele Burden in Patients With JAK2-mutated Myeloproliferative Neoplasms. A Multicenter Phase II Trial.
Brief Title: Sympathicomimetic Agonist in Patients With Myeloproliferative Neoplasms With JAK2-mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 33/14
Record Dates: First submitted 2014-12-04; First posted 2014-12-08 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Myeloproliferative Neoplasm; Primary Myelofibrosis; Essential Thrombocythemia; Polycythemia Vera
Keywords: JAK2; Mirabegron; Primary myelofibrosis; beta-3-mimetic drugs; Myeloproliferative neoplasm; Essential thrombocythemia; Polycythemia vera; Betmiga; JAK2-V617F
MeSH Terms: conditions — Myeloproliferative Disorders; Primary Myelofibrosis; Thrombocythemia, Essential; Polycythemia Vera | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm Mirabegron (Experimental): Mirabegron treatment of at least 24 weeks with an initial dose of 25 mg daily during the first week followed by 50 mg Mirabegron daily during the remaining treatment period.
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — 25 mg daily during the first week followed by 50 mg Mirabegron daily during the remaining treatment period.
  Other Names: Betmiga®

SUMMARY:
The aim of this phase II study is to test a novel concept in the treatment of patients with myeloproliferative neoplasms (MPN), a disease of the bone marrow. With no current cure available, MPN are a group of chronic leukemias (blood cancers) in which patients produce too many blood cells. These increased blood cell numbers cause problems to the patient such as bleedings or thrombosis and some patients may progress to acute leukemia, a life threatening condition. Most MPN patients have a gene mutation called JAK2-V617F. The disease is maintained by mutant MPN stem cells that reside in the bone marrow in specialized locations called "niches". These niches need connections to the nervous system. New findings show that these connections are destroyed by the presence of the mutated MPN stem cells. Research teams found that some drugs (beta3-sympathicomimetics) can restore these damaged niches and at the same time reduce the MPN disease manifestation in a mouse model of MPN. Such sympathicomimetic drugs are already being used to treat patients with asthma or hyperactive bladder. These drugs have shown to have only few side effects. The study tests the effects of the beta-3-sympathicomimetic drug Mirabegron (Betmiga®) on MPN disease in 39 patients that carry a JAK2-V617F mutation. The hypothesis is that Mirabegron will have a beneficial effect on bone marrow niche cells and will thereby improve the disease manifestation in MPN patients. This study should provide a rapid answer whether targeting the nervous system of the niche cells could be useful for patients with MPN and warrants to be tested in larger and more long-term studies.

DETAILED DESCRIPTION:
DISEASE BACKGROUND

Myeloproliferative neoplasms (MPN) are clonal stem cell disorders characterized by aberrant proliferation of the erythroid, megakaryocytic and myeloid lineages. They are associated with decreased survival, thromboembolic complications, hemorrhage and an inherent tendency towards leukemic transformation. About 4-6 of 100'000 residents per year are diagnosed with MPN Currently, MPN are subdivided into three disease entities: polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF). Three genes are frequently mutated in MPN and are implicated to be the phenotypic driver mutations: more than 95% of PV patients carry a somatic JAK2-V617F mutation, while about half of the remaining PV patients (2-3%) display mutations in JAK2 exon 12. Thus, almost all patients with PV have somatic mutations in the JAK2 gene. The mutational profiles of ET and PMF are more diverse: JAK2-V617F is found in 50-60% of the patients, whereas the recently described mutations in calreticulin (CALR) occur in 20-25% of the patients. Between 5-8% of the remaining ET and PMF patients carry mutations in the thrombopoietin receptor (MPL) and in 10-15% of the patient the mutation remains to be determined. Quantitative tests are now available to follow the mutant allele burden of each of the JAK2, CALR and MPL mutant alleles.

THERAPY BACKGROUND

No curative treatment exists for MPN, possibly with the exception of allogeneic hematopoietic stem cell transplantation (HSCT), which is applicable only in a minority of patients. Currently, treatments for MPN are not very effective, or extremely costly. Hydroxyurea has been the standard of care for many decades. A reduction in thrombotic complications can be demonstrated in "high risk" MPN patients (age >60, presence of a previous thrombotic event), but hydroxyurea has no effect on the course of disease (no remission or substantial reduction of the mutant allele burden). Interferon alpha (IFNα) is a promising treatment for early stage PV and is currently being tested in phase III studies. However, IFNα is not always well tolerated and in phase II studies only a proportion of patients showed a substantial response. Ruxolitinib, recently approved for PMF with splenomegaly, is effective in reducing spleen size and improving quality of life, but has little effect on the JAK2-V617F mutant allele burden and has so far not been reported to induce remissions. Allogeneic HSCT is reserved for patients with PMF with a poor prognostic score. These including the recently developed JAK2 inhibitors reduce the symptoms of the disease, but, with the exception of pegylated interferon alpha (peg-IFNα), have little effect on the size of the neoplastic clone and are unable to induce molecular remissions. Thus, the percentage of mutant allele burden in hematopoietic cells does not change much even with successful treatment when considering symptom reduction. It is generally expected that reduction in the size of the malignant clone, as a surrogate marker of treatment success, will have the potential to reduce morbidity and result in prolonged survival of patients.

NOVEL TREATMENT

The beta-3-sympathicomimetic drug Mirabegron is currently available as Betmiga® and indicated to treat hyperactive bladder. It is available as a slow release tablet in a 25 mg and 50 mg formulation. Sympathicomimetic drugs are known to relax the smooth muscle in several areas of the human body and are therefore used for inhalation in patients with asthma or as described for this drug to relax the smooth muscle of the bladder to treat urge incontinence. β3-Adrenoceptors mediate a negative inotropic effect in human ventricular cardiomyocytes, which is opposite to that of β1- and β2-adrenergic receptors. Unlike beta1/2-mimetics, that have significant cardiovascular side effects (including hypertrophy), beta3-mimetics have been reported to protect from hypertrophy and are only associated with some risk of tachycardia and palpitations in some patients.

Sympathicomimetic agonists in patients with JAK2-mutated MPN

RATIONALE FOR PERFORMING THE TRIAL

MPN is initiated and maintained from a mutated hematopoietic stem cell (HSC). The interplay between the MPN HSCs and the stem cell niche is increasingly recognized as crucial for the biology of the disease. Dr. Simon Méndez-Ferrer et al, previously demonstrated that nestin-positive mesenchymal stem cells (nestin+ MSCs) within the bone marrow niche are innervated by sympathetic nerve fibers and are important in regulating normal HSCs. New findings by Dr. Méndez-Ferrer's laboratory show that these nestin+ MSCs are strongly reduced in bone marrow from patients with MPN.

Furthermore, in a mouse model of MPN expressing the human JAK2-V617F mutation, this effect was found to be caused by early glial and sympathetic nerve damage and apoptosis of nestin+ MSCs triggered by the mutant HSCs. In vivo depletion of nestin+ cells accelerated MPN progression. Conversely, MPN phenotype could be reversed by compensating for the sympathetic neuropathy by the treatment with a beta-3-sympathicomimetic drug. Mice with JAK2-V617F driven MPN treated with a beta-3-sympathicomimetic agonist not only restored nestin+ MSCs numbers, but also showed correction of thrombocytosis, neutrophilia, and bone marrow fibrosis, and efficiently reduced mutant hematopoietic progenitor numbers in bone marrow and peripheral blood. Thus, treatments with a beta-3 sympathicomimetic agonist corrected the damage inflicted by the MPN clone on the stem cell niche and led to a dramatic improvement of the MPN phenotype. Therefore, beta-3 sympathicomimetic agonists represent a promising novel therapeutic approach to MPN by targeting the stem cell niche rather than the MPN clone itself.

Considering the widely used and established safety track record of beta-3-sympathicomimetic drugs, a phase II study has been selected to test the concept of a beneficial effect of beta sympathicomimetic activity on bone marrow niche cells and through this effect on the disease manifestation in MPN patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of JAK2-V617F positive ET, PV or PMF at primary diagnosis or pretreated
* JAK2-V617F mutant allele burden > 20% in the peripheral blood at study entry
* Patient must give written informed consent before registration
* WHO performance status 0-2
* Age ≥ 18 years
* Adequate hematological values: neutrophils ≥ 1.5 x 109/L, platelets ≥ 100 x 109/ L
* Adequate hepatic function: bilirubin ≤ 1.5 x ULN, AST/ALT/AP ≤ 2.5 x ULN
* Adequate renal function (calculated creatinine clearance > 50 mL/min, according to the formula of Cockcroft-Gault)
* Women are not breastfeeding. Women with child-bearing potential are using effective contraception, are not pregnant and agree not to become pregnant during participation in the trial and during 28 days thereafter. A negative pregnancy test before inclusion (within 7 days) into the trial is required for all women with child-bearing potential. Men agree not to father a child during participation in the trial and during 28 days thereafter.
* Patient compliance and geographic proximity allow proper staging and follow-up.

Exclusion Criteria:

* Leukemic transformation (>20% blasts in blood, marrow or extramedullary site)
* Diabetic neuropathy
* Severe or uncontrolled cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, history of myocardial infarction within the last twelve months, known cardiac rhythm disturbance including atrial fibrillation or QT prolongation
* Uncontrolled hypertension
* Treatment of ET, PV or PMF with IFNα or treatment of PMF with JAK inhibitors such as ruxolitinib within 3 months prior to trial entry.
* Previous malignancy within 5 years with the exception of adequately treated cervical carcinoma in situ or localized non-melanoma skin cancer.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent or interfering with compliance for oral drug intake.
* Treatment with hematopoietic stem cell transplantation
* Concurrent treatment with cytoreductive drugs, other experimental drugs or other anti-cancer therapy as well as treatment in a clinical trial within 2 months prior to trial entry.
* Any serious underlying medical condition (at the judgment of the investigator), which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes, uncontrolled infection (HIV, Hepatitis B and C).
* Known hypersensitivity to trial drug or hypersensitivity to any other component of the trial drug.
* Any concomitant drugs contraindicated for use with the trial drug according to the approved product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Reduction in the burden of mutated alleles of ≥50% at 24 weeks. | at 24 weeks
  Primary endpoint of the trial is reduction in the burden of mutated alleles of ≥50% at 24 weeks (Red-50@24). Patients are defined as success for this endpoint, if they show a reduction of the JAK2-V617F allelic burden of 50% or more 24 weeks ± 4 weeks after registration when compared to baseline, and if they did not start a new MPN treatment before. All other evaluable patients will be considered as failures for this endpoint.

SECONDARY OUTCOMES:
Reduction in the burden of mutated alleles of ≥50% | at 12 weeks
  Reduction in the burden of mutated alleles of ≥50% at 12 weeks (Red-50@12) defined in the same way as the primary endpoint, but evaluated at 12 weeks ± 4 weeks after registration.
Reduction in the burden of mutated alleles of ≥25% | at 24 weeks
  Reduction in the burden of mutated alleles of ≥25% at 24 weeks (Red-25@24): Patients are defined as success for the Red-25@24 endpoint, if they show a reduction of the Jak2-V617F allelic burden of 25% or more 24 weeks ± 4 weeks after registration when compared to baseline, and if they did not start a new MPN treatment before. All other evaluable patients will be considered as failures for this endpoint.
Reduction in the burden of mutated alleles of ≥25% | at 12 weeks
  Reduction in the burden of mutated alleles of ≥25% at 12 weeks (Red-25@12) defined in the same way as the Red-25@24 endpoint, but evaluated at 12 weeks ± 4 weeks after registration.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob R. Passweg, Prof, Study Chair — University Hospital, Basel, Switzerland; Radek Skoda, Prof, Study Chair — University Hospital, Basel, Switzerland
Locations (11):
- Switzerland (11):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni, Bellinzona
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve, Geneva
  - Centre Hospitalier Universitaire Vaudois CHUV, Lausanne
  - Kantonsspital Liestal, Liestal
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Münsterlingen, Münsterlingen
  - Stadtspital Triemli, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drexler B, Passweg JR, Tzankov A, Bigler M, Theocharides AP, Cantoni N, Keller P, Stussi G, Ruefer A, Benz R, Favre G, Lundberg P, Nienhold R, Fuhrer A, Biaggi C, Manz MG, Bargetzi M, Mendez-Ferrer S, Skoda RC; Swiss Group for Clinical Cancer Research (SAKK). The sympathomimetic agonist mirabegron did not lower JAK2-V617F allele burden, but restored nestin-positive cells and reduced reticulin fibrosis in patients with myeloproliferative neoplasms: results of phase II study SAKK 33/14. Haematologica. 2019 Apr;104(4):710-716. doi: 10.3324/haematol.2018.200014. Epub 2018 Nov 8. PMID 30409796